CLINICAL TRIAL: NCT00635193
Title: A Phase 1/2, Open-Label, Adaptive, Randomized Study of Liposomal Doxorubicin With or Without M200 (Volociximab) for the Treatment of Subjects With Advanced Epithelial Ovarian Cancer or Primary Peritoneal Cancer That Have Relapsed After Prior Therapy With a Platinum/Taxane-Based Chemotherapy
Brief Title: Efficacy and Safety Study of M200(Volociximab in Combination With Liposomal Doxorubicin)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206OC202; 2007-000509-31 (EudraCT Number)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Ovarian Cancer, Primary Peritoneal Cancer
Keywords: Ovarian neoplasms; Angiogenesis inhibitors; Angiogenesis; Volociximab; Ovarian cancer; Antibody; Monoclonals
MeSH Terms: conditions — Ovarian Neoplasms | interventions — volociximab; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Other): Three subjects will be treated with liposomal doxorubicin, 40 mg/m2 q4wk, and volociximab, 7.5 mg/kg qwk
  Interventions: Drug: M200 (Volociximab); Drug: Liposomal Doxorubicin
- Cohort 2 (Other): liposomal doxorubicin, 40 mg/m2 q4wk, and volociximab 15 mg/kg qwk
  Interventions: Drug: Liposomal Doxorubicin; Drug: M200 (Volociximab)
- Group A (Other): liposomal doxorubicin, 40 mg/m2 q4wk
  Interventions: Drug: Liposomal Doxorubicin
- Group B (Other): liposomal doxorubicin, 40 mg/m2 q4wk, and volociximab 15 mg/kg q2wk (or other dose and schedule)
  Interventions: Drug: Liposomal Doxorubicin; Drug: M200 (Volociximab)
- Group C (Other): liposomal doxorubicin, 40 mg/m2 q4wk, and volociximab 15 mg/kg qwk (or other dose and schedule)
  Interventions: Drug: Liposomal Doxorubicin; Drug: M200 (Volociximab)

INTERVENTIONS:
Drug: M200 (Volociximab) — 7.5 mg/kg, IV infusion every week until disease progression
  Arms: Cohort 1
Drug: Liposomal Doxorubicin — 40 mg/m2, IV infustions every 4 weeks until disease progression, the maxium number of doses a subject can receive is 12.
Drug: M200 (Volociximab) — 15 mg/kg, IV infusions every week until disease progression
  Arms: Cohort 2; Group C
Drug: M200 (Volociximab) — 15 mg/kg, IV infustions every other week until disease progression
  Arms: Group B

SUMMARY:
This is an open-label study of liposomal doxorubicin with or without volociximab for the treatment of subjects with advanced epithelial ovarian cancer or primary peritoneal cancer relapsed after prior therapy with Plat/Taxane-based chemo. Volociximab is an anti-angiogenic integrin inhibitor being developed for the treatment of solid tumors. Preclinical data with a surrogate volociximab antibody administered as monotherapy indicate encouraging efficacy in terms of tumor reduction and anti-angiogenic effects in mouse ovarian cancer xenograft models. In clinical studies, volociximab has been evaluated in several solid tumor types, including pancreatic, renal, and melanoma, with many subjects who entered the studies with progressive disease remaining progression-free for several months. In all studies in solid tumors, volociximab has shown a favorable safety profile when administered at 10 mg/kg q2wks and more recently at 15 mg/kg qwk. A study of volociximab in combination with liposomal doxorubicin in subjects with ovarian cancer or primary peritoneal cancer who have relapsed after prior platin/taxane therapies is warranted to further evaluate the drug's efficacy and safety. The investigators have thus far activated stage 2 of this study at 11/25 sites. Worldwide, the study aims to enroll 150 subjects.

DETAILED DESCRIPTION:
This is an open-label study of liposomal doxorubicin with or without volociximab for the treatment of subjects with advanced epithelial ovarian cancer or primary peritoneal cancer relapsed after prior therapy with Plat/Taxane-based chemo. Volociximab is an anti-angiogenic integrin inhibitor being developed for the treatment of solid tumors. Preclinical data with a surrogate volociximab antibody administered as monotherapy indicate encouraging efficacy in terms of tumor reduction and anti-angiogenic effects in mouse ovarian cancer xenograft models. In clinical studies, volociximab has been evaluated in several solid tumor types, including pancreatic, renal, and melanoma, with many subjects who entered the studies with progressive disease remaining progression-free for several months.

ELIGIBILITY:
Inclusion Criteria:

* Females aged >= 18 years old at the time of informed consent.
* Advanced (Stage III or IV) histologically documented epithelial ovarian cancer or primary peritoneal cancer (excluding small, round-cell histologies).
* Recurrent or persistent disease.
* Received no more than 2 prior cancer treatment regimens, at least one of which must have included a platinum/taxane based therapy. If the same regimen is given more than once, it will count as one regimen. If components of a regimen are given more than once using the same schedule, it will count as one regimen.
* At least 1 target lesion to assess response by RECIST criteria. (Tumors within a previously irradiated field are designated as non-target)
* Other protocol-defined inclusion criteria apply.

Exclusion Criteria:

* Subjects taking immunomodulatory agents including, but not limited to, interferons, interleukins, systemic steroids, cyclosporine, tacrolimus, calcineurin inhibitors, chronic low dose methotrexate, or azathioprine. (Use of inhaled or intranasal steroids or oral steroids 10 mg/day prednisone or its equivalent are permitted.)
* Subjects who require treatment with an anti coagulant with the exception of low dose Aspirin® (81 mg/day), warfarin (1 mg/day), or heparin for IV catheter patency
* Evidence of bleeding diathesis or coagulopathy. (Prior history of DVT will not exclude subjects from participating in this study.)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
* Non-healing wound, ulcer, or bone fracture.
* Evidence of autoimmune disease including, but not limited to, ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, scleroderma, and other disease in which immune function or immune competence is known to be impaired.
* Active infection requiring systemic antibiotics, antivirals, or antifungals including HIV/AIDS, hepatitis B, or hepatitis C infection.
* Other protocol-defined exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of volociximab in combination with liposomal doxorubicin in advanced epithelial ovarian cancer or primary peritoneal cancer. To evaluate the safety and tolerability of volociximab in combination with liposomal doxorubicin. | 50-57 days

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — AbbVie
Locations (39):
- United States (14):
  - Site Reference ID/Investigator# 75281, Anaheim, California
  - Site Reference ID/Investigator# 75275, Redondo Beach, California
  - Site Reference ID/Investigator# 75296, Sunrise, Florida
  - Site Reference ID/Investigator# 75299, Atlanta, Georgia
  - Site Reference ID/Investigator# 75300, Savannah, Georgia
  - Site Reference ID/Investigator# 75301, Hinsdale, Illinois
  - Site Reference ID/Investigator# 75274, Baltimore, Maryland
  - Site Reference ID/Investigator# 75294, Jackson, Missouri
  - Site Reference ID/Investigator# 75279, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 75295, Corpus Christi, Texas
  - Site Reference ID/Investigator# 75280, Dallas, Texas
  - Site Reference ID/Investigator# 75297, Danville, Virginia
  - Site Reference ID/Investigator# 75298, Williamsburg, Virginia
  - Site Reference ID/Investigator# 75278, Green Bay, Wisconsin
- Australia (2):
  - Site Reference ID/Investigator# 75334, Toorak Gardens
  - Site Reference ID/Investigator# 75335, Woodville South
- Belgium (3):
  - Site Reference ID/Investigator# 75337, Antwerp
  - Site Reference ID/Investigator# 75336, Brussels
  - Site Reference ID/Investigator# 75338, Leuven
- Italy (2):
  - Site Reference ID/Investigator# 75415, Milan
  - Site Reference ID/Investigator# 75333, Milan
- Poland (7):
  - Site Reference ID/Investigator# 75344, Bialystok
  - Site Reference ID/Investigator# 75339, Krakow
  - Site Reference ID/Investigator# 75341, Lublin
  - Site Reference ID/Investigator# 75342, Poznan
  - Site Reference ID/Investigator# 75343, Poznan
  - Site Reference ID/Investigator# 75345, Szczecin
  - Site Reference ID/Investigator# 75340, Wroclaw
- Russia (3):
  - Site Reference ID/Investigator# 75346, Moscow
  - Site Reference ID/Investigator# 75348, Moscow
  - Site Reference ID/Investigator# 75347, Saint Petersburg
- Spain (5):
  - Site Reference ID/Investigator# 75349, Barcelona
  - Site Reference ID/Investigator# 75351, Barcelona
  - Site Reference ID/Investigator# 75352, Barcelona
  - Site Reference ID/Investigator# 75350, Girona
  - Site Reference ID/Investigator# 75353, Madrid
- Sweden (2):
  - Site Reference ID/Investigator# 75354, Stockholm
  - Site Reference ID/Investigator# 75355, Umeå
- Site Reference ID/Investigator# 75416, Bellinzona, Switzerland

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274